CLINICAL TRIAL: NCT01664117
Title: Study of the Profile and Clinical Management of Patients With Rheumatoid Arthritis Treated With Biologic Therapy Alone
Brief Title: An Observational Study in Clinical Practice Management of Patients With Biological Drugs in Monotherapy
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28356; ROC-BIO-2011-01 (Other: Agencia Española del Medicamento y Productos Sanitarios)
Record Dates: First submitted 2012-08-08; First posted 2012-08-14 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- bDMARD Monotherapy: Patients with moderate to severe rheumatoid arthritis (RA) will be treated with bDMARD (biologic disease-modifying antirheumatic drug) monotherapy under routine clinical practice conditions at rheumatology clinics

SUMMARY:
This observational multicenter study will evaluate the management of disease and safety in clinical practice in patients with moderate to severe rheumatoid arthritis receiving any biological therapies in monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Patients with moderate to severe rheumatoid arthritis who have had an inadequate response or intolerance to disease modifying antirheumatic drugs (DMARDs) or other biological drugs
* Patients treated with biologic DMARDs alone for at least 6 months

Exclusion Criteria:

* Patients not willing or unable to give written informed consent for participation in this study
* Patients who are participating in any clinical trial at the time of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- Spain (36):
  - Vitoria-Gasteiz, Alava
  - Alicante, Alicante
  - Elche, Alicante
  - Zafra, Badajoz
  - Ibiza Town, Balearic Islands
  - Inca, Balearic Islands
  - Manacor (Islas Baleares), Balearic Islands
  - Sabadell, Barcelona
  - Viladecans, Barcelona
  - Burgos, Burgos
  - Cáceres, Caceres
  - Jerez de la Frontera, Cadiz
  - Vinaròs, Castellon
  - Córdoba, Cordoba
  - Girona, Girona
  - Cenes de la Vega, Granada
  - Granda, Granada
  - Donostia / San Sebastian, Guipuzcoa
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - Benalmádena, Malaga
  - Málaga, Malaga
  - Murcia, Murcia
  - Palencia, Palencia
  - Vigo, Pontevedra
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Santa Cruz de Tenerife, Tenerife
  - Toledo, Toledo
  - Gandia, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Zamora, Zamora
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 210 participants were enrolled from 38 rheumatology units in Spain. This study was conducted between June 2012 and June 2013.
Pre-assignment Details: Of 210 participants, one participant was excluded from the study because of past history of biologic disease-modifying antirheumatic drug (bDMARD) monotherapy under 6 months. Therefore, 209 participants were evaluated in this study.
Groups:
- bDMARD Monotherapy: Participants on bDMARD monotherapy for rheumatoid arthritis (RA) in routine clinical practice.
Period: Overall Study
Arm/Group | bDMARD Monotherapy
Started | 209
Completed | 209
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.61 (13.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Level of Education Completed
Description: Level of education completed is a component of socio-demographic characteristics. It is recorded as cannot read, no formal education, primary education or equivalent, general secondary education, vocational education, and higher education or equivalent. Data were collected at study entry (Single visit study)
Time Frame: At Visit 1 (Single visit study)
Population: Analysis population included all enrolled participants who met the screening criteria
Measure: Number; unit: Participants
Groups:
- bDMARD Monotherapy: Participants on bDMARD monotherapy for RA in routine clinical practice.
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Cannot read | 01
  No formal education | 15
  Primary education or equivalent | 86
  General secondary education | 59
  Vocational education | 17
  Higher education or equivalent | 28
  Missing | 03

2. Primary Outcome: Number of Participants With Smoking Habits
Description: Smoking habits is a component of socio-demographic characteristics. Participants' smoking status is recorded as non-smoker, smoker, and ex-smoker at Visit 1.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Non-smoker | 170
  Smoker | 15
  Ex-smoker | 23
  Missing | 01

3. Primary Outcome: Smoking-habit for Smokers or Ex-smokers (Packs in Years)
Description: Smoking-habit included number of pack per years is reported.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria. n = number of evaluated participants
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 38
Years
  Number of pack-years, smoker, n = 15 | 120.20 (138.33)
  Number of pack-years, ex-smoker, n = 23 | 122.26 (122.08)

4. Primary Outcome: Smoking-habit or Smokers or Ex-smokers (Smoking/Quit Smoking )
Description: Smoking-habit included years of smoking/quit smoking is reported for participants.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria. 'n' = number of evaluated participants
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 38
Years
  Years smoking/quit smoking, smoker, n = 15 | 18.73 (9.84)
  Years smoking/quit smoking, ex-smoker, n = 23 | 9.35 (8.39)

5. Primary Outcome: Mean Time of Onset of Rheumatoid Arthritis
Description: Onset of rheumatoid arthritis is a component of clinical characteristics.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Years | 13.45 (8.77)

6. Primary Outcome: Number of Participants With Family History of Rheumatoid Arthritis
Description: Family history is a component of clinical characteristics. Participants who had a family history of rheumatoid arthritis is recorded as yes/no. Also, family history related to parents, siblings, aunts and uncles, grandparents, or other is recorded.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Yes | 15
  No | 160
  Unknown | 34

7. Primary Outcome: Number of Participants With Co-morbidities
Description: Co-morbidity is a component of clinical characteristics It included stroke, heart failure (grades I, II, III or IV), ischemic heart disease, hypertension, dyslipidemia, osteoporosis, interstitial lung disease, chronic obstructive pulmonary disease (COPD), depression, diabetes mellitus, liver disease, serious infections, tuberculosis, hematological malignancies, solid tumors and others. Participants were assessed into categories with associated co-morbidities as yes and no.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Yes | 109
  No | 100

8. Primary Outcome: Number of Participants With Extra-articular Manifestations at Visit 1
Description: Extra-articular manifestations (EAMs) are a component of of clinical characteristics EAMs are symptoms and diseases that occur in parts of the body other than joints. These included the presence of amyloidosis (rare disease that results from the buildup of misfolded proteins), anemia (deficiency of red cells in the blood), heart complications, lung complications, rheumatoid nodules (local swelling), felty's syndrome (presence of rheumatoid arthritis, an enlarged spleen, and an abnormally low white blood cell count), and secondary Sjogren's (an autoimmune disorder that damages moisture-producing glands, making it difficult to produce saliva and tears). Participants were assessed into categories with extra-articular Manifestations as yes, no and missing nos.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Yes | 59
  No | 148
  Missing | 02

9. Primary Outcome: Mean Number of Painful and Swollen Joints at Visit 1
Description: Participants were assessed for painful and swollen joints at Visit 1. Painful joint is the most specific clinical method to quantify abnormalities in participants with RA. It reflects the amount of inflamed synovial tissue.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Number of joints
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Number of joints
  Painful joints | 1.92 (3.00)
  Swollen joints | 0.84 (2.07)

10. Primary Outcome: Physician's Global Assessment of Disease Activity at Visit 1
Description: The Physician's global assessment of disease activity is assessed using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Units on a scale | 2.49 (1.96)

11. Primary Outcome: Patient's Global Assessment of Disease Activity at Visit 1
Description: Patient global assessment of disease activity visual analog scale is assessed using a 0 to 100 mm horizontal VAS. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Units on a scale | 3.11 (2.13)

12. Primary Outcome: Number of Participants With Hematology Parameters Values Falling Within Reference Values at Visit 1
Description: Hematology parameters are considered as one of the component of clinical characteristics. Hematology parameters included white blood cells (WBC), platelets, red blood cells (RBC), hemoglobin, hematocrit, neutrophils, basophils, eosinophils, lymphocytes, monocytes.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria. n =number of evaluated participants
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 192
Participants
  WBC, n = 183 | 159
  Platelets, n = 180 | 165
  RBC, n = 170 | 145
  Hemoglobin, n = 192 | 173
  Haematocrit, n = 174 | 157
  Neutrophils, n = 180 | 140
  Basophils, n = 169 | 164
  Eosinophils, n = 168 | 153
  Lymphocytes, n = 173 | 150
  Monocytes, n = 168 | 152

13. Primary Outcome: Number of Participants With Biochemistry Parameters Values Falling Within Reference Values at Visit 1
Description: Biochemistry parameters is considered as one of the component of clinical characteristics. Biochemistry parameters included alanine amino transferase (ALT), aspartate amino transferase (AST), triglycerides, total cholesterol, high density lipoprotein (HDL), low density lipoprotein (LDL), and total lipids.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria. 'n' =number of evaluated participants
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 184
Participants
  ALT, n = 184 | 172
  AST, n = 172 | 162
  Triglycerides, n = 144 | 130
  Total cholesterol, n = 156 | 104
  HDL, n = 101 | 82
  LDL, n = 102 | 76
  Total lipids, n = 23 | 21

14. Primary Outcome: Number of Participants With Presence/Absence Rheumatoid Factor and Anti-Cyclic Citrullinated Protein Antibodies
Description: Rheumatoid Factor (RF) is the auto antibody directed against Immunoglobulin G and its concentration is observed in human serum or plasma. Anti-Cyclic Citrullinated Protein Antibodies (Anti-CCP) antibodies are auto antibodies (antibodies directed against 1 or more of an individual's own proteins) that are frequently detected in the blood of rheumatoid arthritis participants.
Time Frame: At Visit 1
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  RF - positive for presence | 125
  RF - negative for presence | 42
  RF - not available | 42
  Anti-CCP antibodies - positive for presence | 80
  Anti-CCP antibodies - negative for presence | 35
  Anti-CCP antibodies - not available | 94

15. Primary Outcome: Number of Participants With C-reactive Protein and Erythrocyte Sedimentation Rate Falling Within Reference Values at Visit 1
Description: The test for C-reactive Protein (CRP) is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultra-sensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement. Erythrocyte sedimentation rate (ESR) is a laboratory test that provides a non-specific measure of inflammation. A higher rate is consistent with inflammation.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  CRP | 180
  ESR | 162

16. Primary Outcome: Patient Pain Visual Analog Scale Score at Visit 1
Description: Participants assessed their pain using a 0 to 10 horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 and is described as "no pain" and the right-hand extreme equals 10 as "unbearable pain"
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria. Out of 209 participants, 207 were analysed for patient pain visual analog scale.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 207
Units on a scale | 3.09 (2.14)

17. Primary Outcome: Number of Participants With Joint Damage at Visit 1
Description: Number of participants with joint damage is recorded as yes and no.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Yes | 154
  No | 55

18. Primary Outcome: Mean Score on Disease Activity Score Based on 28-Joints Count at Visit 1
Description: Disease activity score (DAS) 28 is a combined index for measuring disease activity in RA. The index includes swollen (range 0-28) and tender (range 0-28) joint counts, acute phase response (ESR in mm/hr), and general health status (participant global assessment of disease activity using VAS, range 1-100 mm). DAS28, which uses a 28-joint count, is derived from the original DAS, which includes a 44-swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores indicate worsening.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Units on a scale | 2.70 (1.09)

19. Primary Outcome: Number of Participants With Disease Activity Score by Categorization at Visit 1
Description: DAS28 is divided into 4 categories as: remission <2.6, low activity 2.6-3.2, moderate 3.2-5.1 and high >5.1.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Remission | 104
  Low activity | 43
  Moderate activity | 59
  High activity | 03

20. Primary Outcome: Mean Score on Clinical Disease Activity Index at Visit 1
Description: Clinical disease activity index (CDAI) of participants is a composite index that is calculated as the sum of number of painful joint, number of swollen joint, patient's VAS (0-10 cm) assessment, physician global VAS assessment (0-10 cm). The CDAI score ranges from 0 to 76, where lower scores indicate less disease activity.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Scores on a scale | 8.36 (6.94)

21. Primary Outcome: Number of Participants With Clinical Disease Activity by Categorization at Visit 1
Description: CDAI is divided into 4 categories as: remission <2.8, low activity 2.8-10, moderate 10-22 and high>22.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Remission | 33
  Low activity | 118
  Moderate activity | 52
  High activity | 06

22. Primary Outcome: Mean Score on Simple Disease Activity Index at Visit 1
Description: Simple Disease Activity Index (SDAI) is calculated by sum of number of painful joint and swollen joint count, patient and physician global assessment of disease activity (VAS 0-10 cm), and level of C-reactive protein in milligrams per deciliter (mg/dL). SDAI total score ranges from 0 to 86, where higher scores indicates greater affect due to disease activity.
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Scores on a scale | 8.76 (7.06)

23. Primary Outcome: Number of Participants With Simple Disease Activity Index Score by Categorization at Visit 1
Description: SDAI is divided into 4 categories as: remission (<3.3), low activity (3.3-11), moderate activity (11-26) and high activity (>26).
Time Frame: At Visit 1
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Remission | 42
  Low activity | 110
  Moderate activity | 53
  High activity | 04

24. Secondary Outcome: Number of Participants Prescribed First Synthetic Disease-Modifying Antirheumatic Drug Therapy Before the Study
Description: Number of participants prescribed with first synthetic disease-modifying antirheumatic drug therapy (sDMARD) in monotherapy and in a combination before the study was presented.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  First sDMARD as monotherapy | 209
  First sDMARD as combination | 27

25. Secondary Outcome: Mean Time Between Diagnosis and Prescription of First Synthetic Disease-Modifying Antirheumatic Drug or First Biologic Disease-Modifying Antirheumatic Drug
Description: Mean time in months at Visit 1 between diagnosis and prescription of first sDMARD/ first bDMARD was presented.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria. 'n' = number of participants prescribed with first sDMARD or bDMARD.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Months
  sDMARD, n = 209 | 19.53 (52.75)
  bDMARD, n = 126 | 89.81 (86.35)

26. Secondary Outcome: Number of Participants Who Received Each sDMARD Before The Study
Description: Number of participants who previously received sDMARDs before the study in at Visit 1 was reported. sDMARDS included azathioprine, penicillamine, sulfasalazine, hydroxychloroquine, gold salts, chloroquine, leflunomide, ciclosporin, methotrexate, and chlorambucil medications.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Azathioprine | 10
  Penicillamine | 5
  Sulfasalazine | 47
  Hydroxychloroquine | 48
  Gold salts | 48
  Chloroquine | 27
  Leflunomide | 130
  Ciclosporin | 16
  Methotrexate | 197
  Chlorambucil | 1

27. Secondary Outcome: Number of Participants Who Received Last sDMARD Prescribed Before the Study
Description: Number of participants who previously received sDMARDs before the study in at Visit 1 was reported. sDMARDS included azathioprine, penicillamine, sulfasalazine, hydroxychloroquine, gold salts, leflunomide, ciclosporin, methotrexate, and leflunomide + methotrexate.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Azathioprine | 1
  Penicillamine | 1
  Sulfasalazine | 13
  Hydroxychloroquine | 10
  Gold salts | 1
  Leflunomide | 62
  Ciclosporin | 1
  Methotrexate | 119
  Leflunomide + methotrexate | 1

28. Secondary Outcome: Number of Participants Prescribed First bDMARD Before the Study
Description: Number of participants prescribed first bDMARD before the study was presented.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants | 126

29. Secondary Outcome: Number of Participants Who Received Each bDMARD Before the Study
Description: Number of participant who received bDMARD (etanercept, infliximab, golimumab, adalimumab, abatacept, tocilizumab, rituximab) before the study was reported in at Visit 1.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 126
participants
  Etanercept | 58
  Infliximab | 48
  Golimumab | 2
  Adalimumab | 61
  Abatacept | 10
  Tocilizumab | 4
  Rituximab | 16
  Anakinra | 2
  Certolizumab | 2

30. Secondary Outcome: Mean Time Between the Last sDMARD and bDMARD Received at Visit 1
Description: Mean time between the last sDMARD and bDMARD received at Visit 1 was presented in months.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the inclusion criteria. 'n' signifies the number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Months
  sDMARD, n=64 | 9.39 (19.96)
  sDMARD + Biologic agent, n=95 | 1.78 (9.06)
  Monotherapy, n=50 | 36.69 (32.54)

31. Secondary Outcome: Number of Participants With Changing the Previous sDMARD/ bDMARD
Description: Any reasons for changing the previous sDMARD/bDMARD treatment were recorded as lack of efficacy, adverse events, intolerance, clinical improvement and other. There may be more than one reason for changing sDMARD/ bDMARD per participant.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria. 'n' represents the number of participants analyzed at a specified time point.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  sDMARD, Lack of efficacy, n = 209 | 343
  sDMARD, Adverse events, n = 209 | 135
  sDMARD, Intolerance, n = 209 | 25
  sDMARD, Clinical improvement, n = 209 | 7
  sDMARD, Other, n = 209 | 40
  bDMARD, Lack of efficacy, n = 126 | 155
  bDMARD, Adverse events, n = 126 | 38
  bDMARD, Intolerance, n = 126 | 5
  bDMARD, Clinical improvement, n = 126 | 2
  bDMARD, Other, n = 126 | 10

32. Secondary Outcome: Number of sDMARD and bDMARDs Received Before the Study Treatment (bDMARD Monotherapy)
Description: Number of sDMARD and bDMARDs received by Participants before the study was presented
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria. 'n' signifies the number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: Number of sDMARD/bDMARD
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Number of sDMARD/bDMARD
  Number of sDMARD received before the study, n=209 | 2.63 (1.36)
  Number of bDMARD received before the study, n=126 | 1.67 (0.93)

33. Secondary Outcome: Number of Participants Received sDMARD, sDMARD+ bDMARD or bDMARD Immediately Before the Study Treatment
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  sDMARD | 64
  sDMARD+ bDMARD | 95
  bDMARD | 50

34. Secondary Outcome: Number of Participants Discontinued the Previous Treatment and Started the Study Treatment
Description: The reasons for changing the previous sDMARD, sDMARD+ bDMARD or bDMARD treatment and starting the study treatment were recorded as lack of efficacy, adverse events, intolerance, clinical improvement, and other.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Lack of efficacy | 128
  Adverse events | 21
  Intolerance | 16
  Clinical improvement | 22
  Other | 22

35. Secondary Outcome: Median Time Taking the Biologic Agent in Monotherapy Before the Study Treatment
Description: Median time in months taking the Biologic Agent in monotherapy before the study was presented.
Time Frame: At Visit 1
Population: as for outcome 32
Measure: Median (Full Range); unit: Months
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 50
Months
  Etanercept, n = 14 | 29.4 [0.7 to 95.9]
  Infliximab, n = 9 | 31.9 [8.2 to 118.9]
  Golimumab, n = 1 | 59.5 [59.5 to 59.5]
  Adalimumab, n = 15 | 16 [2.0 to 47.9]
  Abatacept, n = 4 | 18.6 [14.3 to 27.6]
  Tocilizumab, n = 1 | 10.1 [10.1 to 10.1]
  Rituximab, n = 6 | 4.1 [0.0 to 34.9]

36. Secondary Outcome: Number of Participants Treated With Concomitant Medications Before the Study
Description: Participants received concomitant medications (corticosteroids, non-steroidal anti-inflammatory drugs [NSAID], and other treatment) before the study were presented.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Corticosteroids | 140
  Non-steroidal anti-inflammatories drugs | 128
  Other treatment | 19

37. Secondary Outcome: Number of Participants Received Current bDMARD Treatment at the Time of the Study
Description: Current bDMARD treatment included etanercept, infliximab, adalimumab, abatacept, tocilizumab, rituximab and certolizumab.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Etanercept | 39
  Infliximab | 3
  Adalimumab | 26
  Abatacept | 8
  Tocilizumab | 122
  Rituximab | 8
  Certolizumab | 3

38. Secondary Outcome: Number of Participants Received Other Concomitant Treatments With the Current bDMARD Monotherapy
Description: Other treatments included corticosteroids, NSAIDs and corticosteroid + NSAID.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Corticosteroids | 39
  NSAID | 48
  Corticosteroid + NSAID | 42

39. Secondary Outcome: Number of Participants With Reasons for Starting Current Biologic Monotherapy
Description: The reasons for changing current biologic treatment were recorded as lack of efficacy, adverse events, intolerance, clinical improvement and other.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Lack of efficacy | 128
  Adverse events | 21
  Intolerance | 22
  Clinical improvement | 22
  Other | 16

40. Secondary Outcome: Number of Participants Who Received Tocilizumab, Anti-Tumour Necrosis Factor and Other as a Monotherapy at the Time of the Study
Description: Participants who received tocilizumab, Anti-tumour necrosis factor (TNF) and Other treatment of monotherapy were reported.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
participants
  Tocilizumab | 122
  ANTI-TNF | 71
  Other | 16

41. Secondary Outcome: Mean Time of bDMARD Monotherapy Started at the Time of the Study Since Onset of RA
Time Frame: At Visit 1
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: years
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
years
  Tocilizumab, n = 122 | 11.34 (7.95)
  Other, n = 87 | 10.23 (9.30)

42. Secondary Outcome: Number of sDMARD and bDMARDs Received Before the Study Treatment (Tocilizumab or Other Biologic Agent)
Time Frame: At Visit 1
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Number of sDMARD/bDMARDs/Other
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Number of sDMARD/bDMARDs/Other
  No. of sDMARDs tocilizumab before the study,n=122 | 2.59 (1.47)
  Other before the study, n=87 | 2.69 (1.20)
  bDMARDs-Tocilizumab before the study,n=122 | 1.34 (1.10)
  bDMARDs-Other before the study, n=87 | 0.53 (0.87)

43. Secondary Outcome: Mean Score on Disease Activity Score Based on 28-Joints Count, Clinical Disease Activity Index and Simple Disease Activity Index by Biologic Agent in Monotherapy at the Time of the Study
Description: Mean score of DAS28 index, CDAI index, and SDAI index were recorded for participants who received biologic agent in monotherapy at the time of the study.
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Tocilizumab: Participants on tocilizumab for RA in routine clinical practice.
- Other Treatments: Participants on Other treatments for RA in routine clinical practice.
Arm/Group | Tocilizumab | Other Treatments
Number analyzed (Participants) | 122 | 87
Units on a scale
  DAS28 | 2.52 (1.06) | 2.97 (1.07)
  CDAI | 8.66 (7.30) | 7.94 (6.42)
  SDAI | 8.94 (7.34) | 8.52 (6.67)

44. Secondary Outcome: Number of Participants With Categorization of Disease Activity Based on Disease Activity Score, Clinical Disease Activity Index Score and Simple Disease Activity Index Score
Description: Mean score of categorization (remission/low activity and moderate/high activity) of DAS28 index, CDAI index, and SDAI index was recorded for participants who received biologic agent in monotherapy at the time of the study .
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | Other Treatments
Number analyzed (Participants) | 122 | 87
participants
  DAS28-Remission/low activity | 90 | 57
  DAS28-Moderate/high activity | 32 | 30
  CDAI- Remission/low activity | 84 | 67
  CDAI- Moderate/high activity | 38 | 20
  SDAI- Remission/low activity | 84 | 68
  SDAI- Moderate/high activity | 38 | 19

45. Secondary Outcome: Mean Number of Joint Count for Painful Joints and Swollen Joints by Biologic Agent in Monotherapy at the Time of the Study
Description: Participants who received biologic agent in monotherapy at the time of the study were assessed for a number of painful joints (NPJ) and swollen joints (NSJ).
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Mean (Standard Deviation); unit: Number of joints
Arm/Group | Tocilizumab | Other Treatments
Number analyzed (Participants) | 122 | 87
Number of joints
  Mean number of NPJ | 2.16 (3.30) | 1.57 (2.51)
  Mean number of NSJ | 0.96 (2.32) | 0.68 (1.65)

46. Secondary Outcome: Number of Participants Falling Within Reference Values For C-reactive Protein and Erythrocyte Sedimentation Rate by Biologic Agent in Monotherapy at the Time of the Study
Description: Participants who received biologic agent in monotherapy at the time of the study were assessed for C-reactive Protein (CRP) and Erythrocyte Sedimentation Rate (ESR).
Time Frame: At Visit 1
Population: Analysis Population included all enrolled participants who met the screening criteria.
Measure: Number; unit: participants
Arm/Group | Tocilizumab | Other Treatments
Number analyzed (Participants) | 122 | 87
participants
  Falling Within Reference Values For CRP | 110 | 70
  Falling Within Reference Values For ESR | 108 | 54

47. Secondary Outcome: Number of Participants With Adverse Events Leading to a Change of Treatment
Description: An Adverse Event was considered as any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Adverse events were collected as a reason for the change to monotherapy.
Time Frame: At the time of change of treatment
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants | 96

48. Secondary Outcome: Number of Participants With Any Adverse Events and Any Serious Adverse Events
Description: An Any Adverse Events (AEs) is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An Serious Adverse Events (SAEs) is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: At the time of change of treatment (to the current treatment)
Population: Analysis population included all enrolled participants who met the screening criteria.
Measure: Number; unit: Participants
Arm/Group | bDMARD Monotherapy
Number analyzed (Participants) | 209
Participants
  Any AEs | 27
  Any SAEs | 07

ADVERSE EVENTS:
Time Frame: At the time of change of treatment (to the current treatment)
Description: Serious adverse events (SAEs) and non-serious AEs reported leading to a change of treatment
Arm/Group | bDMARD Monotherapy
Serious Adverse Events (participants affected / at risk) | 7/209
Other Adverse Events (participants affected / at risk) | 27/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | bDMARD Monotherapy (N=209)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombopenia (Blood and lymphatic system disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 1
Transaminase value increased (Investigations) | 1
Interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | bDMARD Monotherapy (N=209)
Diarrhoea (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Transaminases increased (Investigations) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.